CLINICAL TRIAL: NCT00565318
Title: A Double-Blind Clinical Trial of Benfotiamine Treatment in Diabetic Nephropathy
Brief Title: Benfotiamine in Diabetic Nephropathy
Acronym: Benfo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Isala (Other); Wörwag Pharma GmbH & Co. KG (Unknown); Predictions Network (Unknown)
Responsible Party: Alaa Alkhalaf, M.D, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BENFO-1; NL17390.075.07
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Diabetic Nephropathy
Keywords: Benfotiamine; Diabetes; Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases | interventions — benphothiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Benfotiamine
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benfotiamine — 3x 300 mg film coated tablet daily (900 mg per day). Duration: 12 weeks.
  Other Names: Milgamma® mono 300, Wörwag Pharma GmbH & Co. KG; A11DA05
  Arms: A
Drug: Placebo — 3x 1 film coated tablet daily. Duration: 12 weeks.
  Other Names: Placebo, Wörwag Pharma GmbH & Co. KG
  Arms: B

SUMMARY:
The purpose of this study is to investigate the effect of benfotiamine supplementation in patients with diabetic nephropathy, and to determine whether it will slow down the progression to end-stage renal disease (ESRD).

DETAILED DESCRIPTION:
There is a worldwide increase in prevalence in type 2 diabetes mellitus, which is being paralleled by an increasing number of patients reaching dialysis because of diabetic nephropathy. Much of the fivefold increase in patients receiving dialysis treatment that occurred over the past two decades is attributable to type 2 diabetes and diabetic nephropathy. Diabetes is now the leading cause of end-stage renal disease (ESRD), with more than 40% of all new cases of ESRD occurring in patients with diabetes.

Benfotiamine has been shown to reduce diabetic nephropathy and retinopathy in animal experimental models. We hypothesize that benfothiamine supplementation in patients with diabetic nephropathy will ameliorate the effects of both albuminuria/proteinuria and hyperglycaemia on oxidative stress and advanced glycation end-products (AGEs) accumulation in renal tissue, and thereby decrease inflammatory responses and fibrotic responses, causing slowing down of progression to ESRD as a consequence.

Intervention:

The intervention duration is 12 weeks for each group.

* Group A: Benfotiamine (300 mg) 3x 1 film coated tablet daily (900 mg daily dose benfotiamine)
* Group B: Placebo 3x 1 film coated tablet daily

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Patients are on treatment with angiotensin converting enzyme inhibitors (ACEi) and/or angiotensin II antagonists (AIIA) in an unchanged dose for at least 3 months
* Active diabetic nephropathy as indicated by presence of microalbuminuria (15-300 mg/24 h urine) in at least two samples within 2-6 weeks in advance of inclusion in the trial
* HbA1c < 8.5%, a higher HbA1c < 9.5% is acceptable if the treating physician and the patient have accepted that striving for lower values is an unreachable goal (patients with high HbA1c values are the ones that one would expect to be benefit most from treatment with benfotiamine)
* eGFR (estimated by MDRD formula) > 30 ml/min
* Males and postmenopausal females
* Written informed consent

Exclusion Criteria:

* Renal impairment by other causes than diabetes
* Stage of the disease more severe than indicated in Inclusion criteria (macroalbuminuria or renal insufficiency)
* Severe hypoglycemia during the last 3 months, needing help from another person
* Severe hepatopathy (laboratory values about three times higher than normal
* Endocrine disorders, e.g. hyper/hypothyroidism
* Blood pressure > 160/90 mmHg
* Severe cardiac function disturbances and severe heart rhythm disturbances
* Neoplasm's (excluding history of treated skin cancer of the type basal cell carcinoma BCC or squamous cell carcinoma SCC)
* Severe general diseases or mental disorders making the participation in the study impossible
* Drug abuse
* Female patients during pregnancy and lactation period and female patients with active menses during the past year
* Hypersensitivity to benfotiamine
* HbA1c > 9.5%
* Use of thiamine containing supplements during the last 3 months
* Participation in another study within one month before joining the benfotiamine study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in urinary excretion of: - Kidney injury molecule-1 (KIM-1) - Albumin | 12 weeks

SECONDARY OUTCOMES:
Change in urinary excretion of: β2 microglobulin, macrophage inhibiting factor (MIF), monocyte chemo-attractant protein-1 (MCP-1), and other advanced glycation end-products (AGEs). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: G J Navis, MD, PhD, Study Director — University Medical Center Groningen; H JG Bilo, MD, PhD, Principal Investigator — Isala
Locations (1):
- Isala Klinieken Hospital, Zwolle, Netherlands

REFERENCES:
- [Background] Hammes HP, Du X, Edelstein D, Taguchi T, Matsumura T, Ju Q, Lin J, Bierhaus A, Nawroth P, Hannak D, Neumaier M, Bergfeld R, Giardino I, Brownlee M. Benfotiamine blocks three major pathways of hyperglycemic damage and prevents experimental diabetic retinopathy. Nat Med. 2003 Mar;9(3):294-9. doi: 10.1038/nm834. Epub 2003 Feb 18. PMID 12592403
- [Background] Bakker SJ, Heine RJ, Gans RO. Thiamine may indirectly act as an antioxidant. Diabetologia. 1997 Jun;40(6):741-2. No abstract available. PMID 9222658
- [Background] Thornalley PJ, Babaei-Jadidi R, Al Ali H, Rabbani N, Antonysunil A, Larkin J, Ahmed A, Rayman G, Bodmer CW. High prevalence of low plasma thiamine concentration in diabetes linked to a marker of vascular disease. Diabetologia. 2007 Oct;50(10):2164-70. doi: 10.1007/s00125-007-0771-4. Epub 2007 Aug 4. PMID 17676306
- [Derived] Alkhalaf A, Kleefstra N, Groenier KH, Bilo HJ, Gans RO, Heeringa P, Scheijen JL, Schalkwijk CG, Navis GJ, Bakker SJ. Effect of benfotiamine on advanced glycation endproducts and markers of endothelial dysfunction and inflammation in diabetic nephropathy. PLoS One. 2012;7(7):e40427. doi: 10.1371/journal.pone.0040427. Epub 2012 Jul 6. PMID 22792314
- [Derived] Alkhalaf A, Klooster A, van Oeveren W, Achenbach U, Kleefstra N, Slingerland RJ, Mijnhout GS, Bilo HJ, Gans RO, Navis GJ, Bakker SJ. A double-blind, randomized, placebo-controlled clinical trial on benfotiamine treatment in patients with diabetic nephropathy. Diabetes Care. 2010 Jul;33(7):1598-601. doi: 10.2337/dc09-2241. Epub 2010 Apr 22. PMID 20413516